CLINICAL TRIAL: NCT03905863
Title: A Randomized Controlled Multicentre Trial, Examining the Effect of Natrox® Oxygen Wound Therapy on the Healing Rate of Chronic Diabetic Foot Ulcers
Brief Title: The Effect of Natrox® Oxygen Wound Therapy on the Healing Rate of Chronic Diabetic Foot Ulcers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inotec AMD Limited (Industry)
Collaborators: SerenaGroup, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Results first posted 2021-11-22 (Actual); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Diabetic Foot Ulcer; Surgical Wound
Keywords: topical oxygen; topical oxygen treatment; diabetic foot ulcer; non-healing wound; surgical site; pain; wound size; healing; infection
MeSH Terms: conditions — Diabetic Foot; Surgical Wound; Pain; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard of care arm (No Intervention): SOC was defined to include wound cleansing with sterile water or saline solution, and gentle irrigation of the study ulcer with warm tap water; sharp debridement using a standardised protocol based on TIME principles for wound bed preparation; offloading with a TCC twice in the first week and weekly thereafter (all exceptions had to be agreed by the lead investigator; a fixed ankle walker boot or similar device was acceptable as an alternative, but shoe inserts were not deemed to provide sufficient offloading); moisture balance was provided using a hydrofibre or alginate dressing. In addition, patients were instructed on adherence to the protocol and given instructions to call their clinic if they suspected any signs of an infection.
- Intervention arm (Active Comparator): Same protocol as SOC only but were also provided with a Natrox® Oxygen Wound Therapy System, consisting of two elements: the Natrox® OG and the Natrox® ODS. The OG is a multi-use battery powered device which generates oxygen though water electrolysis at a rate of 15mL/hr. The ODS is a sterile, single use device that allows wound exudate to pass through to the secondary dressing while allowing the diffusion of oxygen across the wound bed. It connects directly to the OG via a thin flexible fine-bore tube. While the ODS can remain in situ for 7 days, it should be changed at each dressing change, based on exudate level or clinical judgement. This is a battery-operated system with a 30-hour battery life; the kit includes two interchangeable, rechargeable batteries. Each participant was advised to charge one battery while the other was in use, as the battery required changing daily. The oxygen generator is worn in a holster so that patients can remain ambulatory.
  Interventions: Device: Natrox® Oxygen Wound Therapy

INTERVENTIONS:
Device: Natrox® Oxygen Wound Therapy — A battery-operated device which delivers pure humidified oxygen to the wound bed through water electrolysis via a sterile oxygen delivery system.
  Arms: Intervention arm

SUMMARY:
A Multicentre Randomized Controlled Trial to Investigate the Effect of Natrox Topical Oxygen Wound Therapy on the Healing rates of Diabetic Foot Ulcers.

DETAILED DESCRIPTION:
Patients with diabetic foot ulcers will be enrolled into the trial at multiple wound care centers and hospital research centers across the United States of America. After qualifying per protocol, patients will be randomized to receive standard wound care or standard wound care plus Topical Oxygen Wound Therapy for their wounds. Patients will be monitored for 12 weeks. The primary comparator between the groups will be complete wound healing at 12 weeks, but other parameters will be assessed, such as pain, wound size reduction and infection status.

ELIGIBILITY:
Inclusion Criteria

1. Subjects are male or female, 18 years of age or older. At least 50% of the enrolled population must be ≥ 65 years of age.
2. Subjects with one of the following wounds:

   A. Diabetic foot ulcer present for greater than 4 weeks (documented in the medical record) but less than 12 months duration if being treated with active SOC.

   B. Minor amputation wound sites
3. Subject has clinical documentation of no visible wound improvement in the after 4 weeks of standard of care. Objectively, less than 40% healing in the past four weeks from the first treatment visit.
4. Study ulcer is a minimum of 0.5 cm2 and a maximum of 25 cm2 at first treatment visit
5. Subjects' wound score on ISDA tool is Grade 1 or 2.
6. The subject is able and willing to follow the protocol requirements
7. Subject has signed informed consent
8. Adequate circulation to the affected foot as demonstrated by a dorsum transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg; an ABI between 0.7 and ≤ 1.3, or TBI of >6 within 3 months of the first Screening Visit.
9. Females of childbearing potential must be willing to use acceptable methods of contraception (birth control pills, barriers, or abstinence).
10. The target ulcer has been offloaded for at least 14 days prior to randomization.

Exclusion Criteria

1. Subject has a known life expectancy of < 1 year
2. Subject or caregiver is unable to manage the Natrox® device (charge and change batteries daily)
3. Subject has ulcers that are completely necrotic or if the clinician feels it is clinically necessary to cover the wound surface in gel or creams that would prevent the transmission of oxygen to the wound surface.
4. Subject has major uncontrolled medical disorders such as serious cardiovascular, renal, liver or pulmonary disease, lupus, palliative care or sickle cell anemia.
5. Subject currently being treated for an active malignant disease or subjects with history of malignancy within the wound.
6. The Subject has other concurrent conditions that in the opinion of the Investigator may compromise subject safety
7. Known contraindications for the Natrox system
8. Known allergies to any of the Natrox system components
9. Concurrent participation in another clinical trial that involves an investigational drug or device that would interfere with this study.
10. Index ulcer has reduced in area by 20% or more after 2 weeks of standard of care from the first screening visit (S1) to the TV1/randomization visit.
11. Subject is pregnant or breast feeding.
12. Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids >10mg daily dose), cytotoxic chemotherapy, or application of topical steroids to the ulcer surface within one month prior to first Screening Visit, or who receive such medications during the screening period, or who are anticipated to require such medications during the course of the study.
13. Index ulcer has been previously treated with tissue engineered materials (e.g. Apligraf® or Dermagraft®) or other scaffold materials (e.g. Oasis, Matristem) within the last 30 days preceding the first treatment visit.
14. Affected extremity requiring hyperbaric oxygen during the trial or within 2 weeks of treatment visit 1.
15. Known HbA1C >12%
16. An ulcer that has visible signs of improvement in the four weeks prior to randomization defined objectively as a 40% reduction in surface area in the four weeks prior to enrollment.
17. An ulcer that has healed by more than 20% in the 2 weeks prior to screening: "historical" run-in period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2019-06-04 (Actual); Primary Completion 2020-10-18 (Actual); Study Completion 2020-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Serena, Study Director — SerenaGroup, Inc.
Locations (20):
- United States (19):
  - New Hope Podiatry Clinic, Los Angeles, California
  - MedCare Research, Miami, Florida
  - San Marcus Research Clinic, Miami Lakes, Florida
  - Global Health Research Center Inc, Miami Lakes, Florida
  - Barry University Clinical Research, North Miami Beach, Florida
  - Royal Research Corp, Pembroke Pines, Florida
  - Doctors Research Network, South Miami, Florida
  - Pharma Research Associates, Westchester, Florida
  - Wahab Consulting and Research, Las Vegas, Nevada
  - Cleveland Foot and Ankle Clinic, Cleveland, Ohio
  - Tulsa Bone and Joint, Tulsa, Oklahoma
  - The Foot and Ankle Wellness Center of Western Pennsylvania, Ford City, Pennsylvania
  - Antria, Indiana, Pennsylvania
  - ACMH Snyder Institute, Kittanning, Pennsylvania
  - SerenaGroup Research Institute, Pittsburgh, Pennsylvania
  - El Campo Memorial Hospital, El Campo, Texas
  - Allure Health LLC, Friendswood, Texas
  - Pinnacle Foot and Ankle Center, Houston, Texas
  - Mercury Clinical Research, Webster, Texas
- Clinical Research Management Group, Coto Laurel, Ponce, Puerto Rico

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were initially screened and documentation was investigated. If all inclusion criteria were met, and the patient had a documented healing rate of <20% reduction in wound size, the patients were entered into the 2-week run-in period. All patients were allocated to standard of care (SOC). At the baseline visit, if all inclusion and exclusion criteria were still applicable and the wound had not reduced in size by >20%, the patient was then randomized.
Pre-assignment Details: During run-in period patients either exceeded the percentage of acceptable healing per the protocol or had an adverse event preventing continuation in the trial.
Groups:
- Standard of Care Arm: SOC was defined to include wound cleansing with sterile water or saline solution, and gentle irrigation of the study ulcer with warm tap water; sharp debridement using a standardized protocol based on TIME principles for wound bed preparation; offloading with a TCC twice in the first week and weekly thereafter (all exceptions had to be agreed by the lead investigator; a fixed ankle walker boot or similar device was acceptable as an alternative, but shoe inserts were not deemed to provide sufficient offloading); moisture balance was provided using a hydrofibre or alginate dressing. In addition, patients were instructed on adherence to the protocol and given instructions to call their clinic if they suspected any signs of an infection.
- Intervention Arm: Those subjects allocated to the intervention arm were treated using the same protocol as SOC only but were also provided with a Natrox® Oxygen Wound Therapy System, consisting of two elements: the Natrox® Oxygen Generator and the Natrox® Oxygen Delivery System. The oxygen generator is a multi-use battery powered device which generates oxygen though water electrolysis at a rate of 15mL/hr. The oxygen delivery system is a sterile, single use device which has a web-like design that allows wound exudate to pass through to the secondary dressing while allowing the diffusion of oxygen across the wound bed. It connects directly to the oxygen generator via a thin flexible fine-bore tube. While the oxygen delivery device can remain in situ for 7 days, it should be changed at each dressing change, based on exudate level or clinical judgement. This is a battery-operated system with a 30-hour battery life; the kit includes two interchangeable, rechargeable batteries. Each participant was advised to charge one battery while the other was in use, as the battery required changing daily. The oxygen generator is worn in a holster so that patients can remain ambulatory.
Period: Overall Study
Arm/Group | Standard of Care Arm | Intervention Arm
Started | 64 | 81
Completed | 59 | 69
Not Completed | 5 | 12
Not completed — Adverse Event | 2 | 4
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 0 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — Protocol Violation | 0 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Arm: Patients in the standard of care arm will receive the standard care for their type of wound from their wound care centre.
- Intervention Arm: Patients in the intervention arm will receive standard of care plus Natrox® Oxygen Wound Therapy as treatment for their wound.
  Natrox® Oxygen Wound Therapy: A battery-operated device which delivers 98% pure humidified oxygen to the wound bed through water electrolysis via a sterile oxygen delivery system.
- Total: Total of all reporting groups
Arm/Group | Standard of Care Arm | Intervention Arm | Total
Number analyzed (Participants) | 64 | 81 | 145
Age, Continuous [Mean (Full Range); unit: years] | 62.69 [34 to 91] | 64.2 [33 to 93] | 63 [33 to 93]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One patient did not declare.
  Participants
    number analyzed (Participants) | 64 | 80 | 144
    Female | 11 | 26 | 37
    Male | 53 | 54 | 107
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 8 | 5 | 13
  United States | 56 | 76 | 132
Current use Tobacco [Count of Participants; unit: Participants]
  Yes | 11 | 11 | 22
  No | 51 | 68 | 119
  Not declared | 2 | 2 | 4
Diabetes duration [Mean (Full Range); unit: years] — Missing data for 4 patients in Standard of Care and 5 patients in Standard of Care plus Topical Oxygen Therapy. Population: Analysis was only completed on the 2 individual study arms.
  years
    number analyzed (Participants) | 60 | 76 | 136
    (all) | 18.33 [3 to 62] | 18.35 [1 to 55] | 18.34 [1 to 62]
BMI [Mean (Full Range); unit: Kg/m^2] — Missing data on 4 patients in SOC and 5 patients in SOC plus TOT. Population: BMI Analysis: Was only completed on the 2 individual arms.
  Kg/m^2
    number analyzed (Participants) | 60 | 76 | 136
    (all) | 31 [19 to 51] | 30.8 [16 to 54] | 30.9 [16 to 54]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants That Achieve Complete Wound Closure During the Twelve Week Study and the Percentage Change in Participant Ulcer Size at 12 Weeks From Baseline.
Description: Photographic wound evaluation and measurements were conducted utilizing an AI-driven computerized planimetry imaging system (Tissue Analytics, Inc., Baltimore, MD USA).15 This system obtained both 2D and 3D assessments of the wound at each visit through a standardized mobile device; in addition, the lead investigator reviewed all digital images.
Time Frame: Twelve (12) weeks from Time 0
Population: Intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Standard of Care Arm | Intervention Arm
Number analyzed (Participants) | 64 | 81
Participants
  Intention to treat-healed | 18 | 36
  Per protocol-healed: number analyzed (Participants) | 59 | 69
  Per protocol-healed | 18 | 36

2. Primary Outcome: Percentage Reduction in Ulcer Area (cm^2).
Description: Wound size change over time using a wound imaging measurement system. Percentage change in ulcer area was calculated on the basis of area change from the start of the study to the final recorded value. Any healed ulcer was recorded as having achieved 100% reduction in area; positive values indicate a reduction in size over the 12-week period while negative values indicate that the ulcer increased in size.
Time Frame: Twelve (12) weeks from Time 0
Population: "Intention to treat" as well an "Per protocol" analysis was carried out.
Measure: Mean (Standard Deviation); unit: Percentage reduction
Arm/Group | Standard of Care Arm | Intervention Arm
Number analyzed (Participants) | 64 | 81
Percentage reduction
  Intention to treat - percentage reduction | 41.05 (69.82) | 46.38 (100.24)
  Per protocol-percentage reduction: number analyzed (Participants) | 59 | 69
  Per protocol-percentage reduction | 40.44 (72.1) | 70.18 (45.5)

3. Secondary Outcome: Level of Pain of the Wound
Description: Does pain associated with the wound change over time using a Visual Analogue Scale Pain intensity of the reference DFU is to be assessed before any dressing changes or other ulcer manipulations at all screening and treatment visits.
  Subject will be asked to indicate a numerical value that best represents the pain intensity at ulcer site on a scale of 0 to 10 anchored by word descriptors at each end, as "no pain" on the left side and "worst possible pain" on the right side of the number line. The number 0 represent "no pain", the number 5 represents "moderate pain" and the number 10 represents the "worst possible pain". The subject indicates the level of pain intensity by selecting a number on the line that represents their perception of their current state.
Time Frame: Up to twelve (12) weeks from Time 0
Population: VAS scores were taken weekly. On a scale of 0-10, 0 is least pain and 10 is the most pain
Measure: Mean (Standard Deviation); unit: score on a VAS 0-10 scale
Arm/Group | Standard of Care Arm | Intervention Arm
Number analyzed (Participants) | 64 | 81
score on a VAS 0-10 scale
  Baseline | 2.02 (2.57) | 1.81 (2.53)
  Twelve weeks of final visit if healed during study | 0.68 (1.43) | 0.95 (1.9)

4. Secondary Outcome: Number of Adverse Events
Description: Number of adverse events, such as infections, that are found associated with the study wound
Time Frame: Up to twelve (12) weeks from time 0
Population: Adverse reactions were recorded and reported throughout the study as they occurred.
Measure: Number; unit: Number of adverse events
Arm/Group | Standard of Care Arm | Intervention Arm
Number analyzed (Participants) | 64 | 81
Number of adverse events
  Number of adverse events | 32 | 41
  Relationship to the product/unrelated | 30 | 37
  Relationship to the product/Unlikely | 1 | 2
  Relationship to the product/ Possibly related | 1 | 1
  Relationship to the product/ probably related | 0 | 1

ADVERSE EVENTS:
Time Frame: During the12 week intervention period patients were monitored for adverse events.
Description: * Severity of adverse events: Mild, Moderate, Severe, Life Threatening.
  * Outcome: Recovered, Recovered with sequelae, Not recovered, Lost to follow-up, Death.
  * Relationship to product: Unrelated, Unlikely, Possibly related, Probably related.
  * Action taken: Continued, Interrupted time in study, Discontinued.
Groups:
- Standard of Care Arm: Patients in the standard of care arm will receive the standard care for their type of wound from their wound care centre which typically includes a primary and secondary dressing to the wound.
- Intervention Arm: Patients in the intervention arm will receive standard of care plus Natrox® Oxygen Wound Therapy as treatment for their wound.
  Natrox® Oxygen Wound Therapy: A battery-operated device which delivers pure humidified oxygen to the wound bed through water electrolysis via a sterile oxygen delivery system.
Arm/Group | Standard of Care Arm | Intervention Arm
All-Cause Mortality (participants affected / at risk) | 0/64 | 1/81
Serious Adverse Events (participants affected / at risk) | 8/64 | 6/81
Other Adverse Events (participants affected / at risk) | 13/64 | 19/81
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Arm (N=64) | Intervention Arm (N=81)
Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Gangrene (Infections and infestations) | 1 (1) | 1 (1)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Bacteremia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) — Linked to cellulitis previously recorded as an AE
Osteomyelitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0)
Acute hypokalemic (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Associated hypotension and nonischemic cardiomyopathy
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Arm (N=64) | Intervention Arm (N=81)
New Wound (Skin and subcutaneous tissue disorders) | 7 (8) | 6 (6)
Falls (Injury, poisoning and procedural complications) | 2 (2) | 4 (7)
Maceration (Skin and subcutaneous tissue disorders) | 2 (4) | 2 (2)
Wound Infection (Infections and infestations) | 2 (2) | 6 (6)
Infections (Infections and infestations) | 3 (4) | 1 (1)
Pain (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — Wound/leg pain

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2019-11-25): https://cdn.clinicaltrials.gov/large-docs/63/NCT03905863/Prot_SAP_ICF_001.pdf